CLINICAL TRIAL: NCT04069221
Title: An Open-label, Two-part Study to Determine the Absolute Bioavailability (BA) of OZ439 Using Simultaneous Intravenous [14C]-OZ439 Microdose/800mg Oral Dosing and to Investigate the Pharmacokinetics (PK) of OZ439 Granules Administered as Single Doses Suspended in Different Volumes and When Co-administered With a Single Dose of Cobicistat, a Strong CYP3A4 Inhibitor, to Healthy Subjects in Fasted State
Brief Title: Absolute BA and OZ439 PK Effect of Different OZ439 Dose Volumes and Cobicistat Co-administration Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MMV_OZ439_16_01
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — artefenomel

STUDY DESIGN:
Intervention Model Description: Part1: Open label, one treatment Part 2: Open-label, randomized, single-dose, 3-way cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1, single arm (Experimental): This was an open-label study in 8 healthy subjects to determine the absolute bioavailability of OZ439 following a single oral dose of OZ439 and co-administration of a single iv infusion of a [14C]-OZ439 radiolabeled microdose at the anticipated Tmax of the oral dose. Subjects received the following treatment:
  Treatment A: A single oral dose of 800 mg OZ439 simple granules administered as a 100-mL dispersion followed by a 15-minute 10-mL iv infusion of 100 μg [14C]-OZ439 (47 kBq [1.27 μCi]) beginning 3 hours after the oral dose administration.
  Interventions: Drug: Single oral dose of 800 mg OZ439; Drug: iv infusion of [14C]-OZ439
- Part 2, Treatment B: single oral dose of 800 mg OZ439 (Experimental): This was an open-label, randomized, single-dose, 3-way cross-over study in 18 healthy subjects. Each subject participated in 3 treatment periods and each subject received a single dose of each of the following 3 treatments in a randomized order with a 14-day wash-out period between each treatment: Treatment B: A single oral dose of 800 mg OZ439 simple granules administered as a 64.5-mL dispersion Treatment C: A single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion Treatment D: A single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion and co-administered with a 150 mg cobicistat tablet (CYP3A4 inhibitor)
  Interventions: Drug: Single oral dose of 800 mg OZ439
- Part 2, Treatment C: single oral dose of 400 mg OZ439 (Experimental): This was an open-label, randomized, single-dose, 3-way cross-over study in 18 healthy subjects. Each subject participated in 3 treatment periods and each subject received a single dose of each of the following 3 treatments in a randomized order with a 14-day wash-out period between each treatment: Treatment B: A single oral dose of 800 mg OZ439 simple granules administered as a 64.5-mL dispersion Treatment C: A single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion Treatment D: A single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion and co-administered with a 150 mg cobicistat tablet (CYP3A4 inhibitor)
  Interventions: Drug: Single oral dose of 400 mg OZ439
- Part 2, Treatment D:single oral dose 400 mg OZ439+cobicistat (Experimental): This was an open-label, randomized, single-dose, 3-way cross-over study in 18 healthy subjects. Each subject participated in 3 treatment periods and each subject received a single dose of each of the following 3 treatments in a randomized order with a 14-day wash-out period between each treatment: Treatment B: A single oral dose of 800 mg OZ439 simple granules administered as a 64.5-mL dispersion Treatment C: A single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion Treatment D: A single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion and co-administered with a 150 mg cobicistat tablet (CYP3A4 inhibitor)
  Interventions: Drug: Single oral dose of 400 mg OZ439; Drug: Single oral dose of cobicistat

INTERVENTIONS:
Drug: Single oral dose of 800 mg OZ439 — Single oral dose of 800 mg OZ439
  Arms: Part 1, single arm; Part 2, Treatment B: single oral dose of 800 mg OZ439
Drug: Single oral dose of 400 mg OZ439 — Single oral dose of 400 mg OZ439
  Arms: Part 2, Treatment C: single oral dose of 400 mg OZ439; Part 2, Treatment D:single oral dose 400 mg OZ439+cobicistat
Drug: Single oral dose of cobicistat — Single oral dose of 150 mg cobicistat
  Arms: Part 2, Treatment D:single oral dose 400 mg OZ439+cobicistat
Drug: iv infusion of [14C]-OZ439 — 15-minute 10-mL iv infusion of 100 μg [14C]-OZ439
  Arms: Part 1, single arm

SUMMARY:
This study is an open-label, two-part study to determine the absolute bioavailability (BA) of OZ439 using simultaneous intravenous [14C]-OZ439 microdose/800mg oral dosing and to investigate the pharmacokinetics (PK) of OZ439 granules administered as single doses suspended in different volumes and when co-administered with a single dose of Cobicistat, a strong CYP3A4 inhibitor, to healthy subjects in fasted state.

DETAILED DESCRIPTION:
Primary objectives of this study are:

* to determine the absolute bioavailability of OZ439 following a single oral dose of OZ439 dispersion and a simultaneous single intravenous (iv) microdose (100 μg) infusion of [14C]-OZ439 under fasted conditions (Part 1)
* To evaluate the effects of a single oral dose of cobicistat, a strong cytochrome P450 (CYP) 3A4 inhibitor, on the pharmacokinetic (PK) profile of a single oral dose of a dispersion of OZ439 simple granules under fasted conditions (Part 2)
* To evaluate the PK of single doses of OZ439 granules when restricting the target dosing volumes to 64.5 or 100 mL (Parts 1 and 2)

Secondary objectives are:

* To assess the safety and tolerability of OZ439 when administered alone, and to assess the safety and tolerability of OZ439 and cobicistat when co-administered as single doses to healthy subjects (Parts 1 and 2)
* To determine the PK parameters of OZ439 single iv microdose (100 μg) infusion of [14C]-OZ439 (Part 1)
* To assess the effects of the total dosing volume and of dose to volume ratio on OZ439 PK under fasted conditions (Parts 1 and 2)
* To determine the PK parameters and exposures of cobicistat (Part 2)

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) : 18.0-30.0 kg/m2, inclusive, at screening
* Weight : >50 kg, at screening
* Status : healthy subjects
* Female subjects must be of non-childbearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or post-menopausal [defined as spontaneous amenorrhoea for at least 1 year or spontaneous amenorrhoea for at least 6 months confirmed by a follicle stimulating hormone (FSH) result indicating a post-menopausal status]) and have a negative pregnancy test at screening and at (each) admission to the clinical research center. As all female subjects must be of non-childbearing potential, they are not required to use any contraception during this study.
* Male subjects must use adequate contraception and not donate sperm from (first) admission to the clinical research center until 90 days after the follow-up visit. Adequate contraception for the male subject (and his female partner) is defined as surgical sterilization (vasectomy), using hormonal contraceptives (implantable, patch, oral, injectable) or an intrauterine device or system combined with at least 1 of the following forms of contraception (barrier method): a diaphragm or cervical cap, or a condom. Also, total abstinence, in accordance with the lifestyle of the subject is acceptable.
* Must have QTcF ≤450 ms and QTcB ≤450 ms (male subjects); QTcF ≤470 ms and QTcB ≤470 ms (female subjects), and PR-interval ≤200 ms for screening, and Day -1 and pre-dose ECG measurements of the (first) treatment period
* Ability and willingness to abstain from alcohol and methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks) from 48 hours prior to (each) admission to the clinical research center
* Willing and able to communicate and participate in the whole study
* Willing and able to sign the ICF

Exclusion Criteria:

* A subject who meets any of the following exclusion criteria will not be eligible for inclusion in the study:
* Male subjects who have currently pregnant partners or who have partners planning to be pregnant in the 90 days after discharge
* Evidence or history of clinically significant oncological, pulmonary, chronic respiratory, hepatic, cardiovascular, hematological, metabolic, neurological, immunological, nephrological, endocrine or psychiatric disease, or current infection
* Clinically relevant (as decided by the Principal Investigator [PI]) abnormalities in the 12-lead ECG, including asymptomatic bundle branch block
* Family history of sudden death or of congenital prolongation of the QTc-interval or known congenital prolongation of the QTc-interval or any clinical condition known to prolong the QTc-interval
* History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia, heart rate ≤39 beats per minute (bpm)
* Electrolyte disturbances, particularly hypokalemia, hypocalcemia or hypomagnesemia
* Any condition that could possibly affect drug absorption, e.g. gastrectomy or diarrhea
* History of post-antibiotic colitis
* History of any drug or alcohol abuse in the past 2 years prior to screening
* Subjects who regularly smoke more than 5 cigarettes a day
* Receipt of an investigational drug or participation in another clinical research study within 90 days prior to the first dose of study drug
* Subjects who are PRA employees, or immediate family members of PRA or Sponsor employees
* Subjects who have previously been enrolled in this study
* Use of moderate/strong inhibitors or inducers of CYP cytochromes or transporters within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug
* Consumption of grapefruit, grapefruit juice or grapefruit-related citrus fruits (e.g. Seville oranges, pomelos) within 14 days prior to the first dose of study drug
* Use of prescription or non-prescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study drug. With the exception of paracetamol (which may be used incidentally or for a short-term treatment at a maximum dose of 2 g per day) and hormone replacement therapy
* Use of herbal supplements within 30 days prior to the first dose of study drug
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or HIV-1 or HIV-2 antibody results
* Clinically significant abnormal biochemistry, hematology or urinalysis as judged by the PI. In case of doubt the PI will discuss this with the medical monitor
* Positive urine drug screen result at screening or admission to the clinical research center
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of allergy requiring treatment. Hayfever is allowed unless it is active
* Donation or loss of >100 mL of blood within 90 days prior to drug administration
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = 250 mL beer, 25 mL of 40% spirit or 125 mL of wine)
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the PI or delegate at screening
* Failure to satisfy the PI of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences (PRA) - Early Development Services (EDS), Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screened volunteers: 48
  Screening failures:
  ECG: 7 Clinical laboratory: 3 Medical history: 2 Vital signs: 1 Physical examination: 1 Other: 1
  Approved but not dosed Reserve: 5 Not in clinic/Personal: 2
Groups:
- Part 1: open-label study in 8 healthy subjects to determine the absolute bioavailability of OZ439 following a single oral dose of OZ439 and co-administration of a single iv infusion of a [14C] OZ439 radiolabeled microdose
- Part 2 Treatment B, Then C and D: open-label, randomized, single-dose, 3-way cross-over study in 18 healthy subjects. Each subject participated in 3 treatment periods and each subject received a single dose of each of the following 3 treatments in a randomized order with a 14-day wash-out period between each treatment
  * Treatment B: a single oral dose of 800 mg OZ439 simple granules administered as a 64.5-mL dispersion
  * Treatment C: a single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion
  * Treatment D: a single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion and co-administered with a 150 mg cobicistat tablet (CYP3A4 inhibitor)
- Part 2 Treatment C, Then D and B: open-label, randomized, single-dose, 3-way cross-over study in 18 healthy subjects. Each subject participated in 3 treatment periods and each subject received a single dose of each of the following 3 treatments in a randomized order with a 14-day wash-out period between each treatment
  * Treatment C: a single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion
  * Treatment D: a single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion and co-administered with a 150 mg cobicistat tablet (CYP3A4 inhibitor)
  * Treatment B: a single oral dose of 800 mg OZ439 simple granules administered as a 64.5-mL dispersion
- Part 2 Treatment D, Then B and C: open-label, randomized, single-dose, 3-way cross-over study in 18 healthy subjects. Each subject participated in 3 treatment periods and each subject received a single dose of each of the following 3 treatments in a randomized order with a 14-day wash-out period between each treatment
  * Treatment D: a single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion and co-administered with a 150 mg cobicistat tablet (CYP3A4 inhibitor)
  * Treatment B: a single oral dose of 800 mg OZ439 simple granules administered as a 64.5-mL dispersion
  * Treatment C: a single oral dose of 400 mg OZ439 simple granules administered as a 64.5-mL dispersion
Period: Overall Study
Arm/Group | Part 1 | Part 2 Treatment B, Then C and D | Part 2 Treatment C, Then D and B | Part 2 Treatment D, Then B and C
Started | 8 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 2: open-label, randomized, single-dose, 3-way cross-over study in 18 healthy subjects. Each subject participated in 3 treatment periods and each subject received a single dose of each of the following 3 treatments in a randomized order with a 14-day wash-out period between each treatment
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 8 | 18 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 18 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 18 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Black | 1 | 0 | 1
  White | 5 | 15 | 20
  Hispano or Latino | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: OZ439 Fpo
Description: OZ439 Absolute oral bioavailability
Time Frame: OZ439: Pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 168 hours post-dose. [14C]-OZ439: 10, 15, 20, 30 and 45 minutes after start of iv infusion then 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 168 hours
Measure: Geometric Mean (90% Confidence Interval); unit: Absolute bioavailability in %
Groups:
- Part 1: open-label study in 8 healthy subjects to determine the absolute bioavailability of OZ439 following a single oral dose of OZ439 and co-administration of a single iv infusion of a [14C] OZ439 radiolabeled microdose at the anticipated tmax of the oral dose.
  Treatment A: a single oral dose of 800 mg OZ439 simple granules administered as a 100-mL dispersion followed by a 15-minute 10-mL iv infusion of 100 μg [14C] OZ439 (47 kBq [1.27 µCi]) beginning 3 hours after the oral dose administration.
Arm/Group | Part 1
Number analyzed (Participants) | 8
Absolute bioavailability in % | 35 [29 to 41]

2. Primary Outcome: OZ439 Cmax
Description: OZ439 maximum concentration observed
Time Frame: Pre-dose, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 168, 216, 264, 312 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2, Treatment B: Single Oral Dose of 800 mg OZ439 | Part 2, Treatment C: Single Oral Dose of 400 mg OZ439 | Part 2, Treatment D:Single Oral Dose 400 mg OZ439+Cobicistat
Number analyzed (Participants) | 18 | 18 | 18
ng/mL | 949 (36.1) | 649 (40.7) | 966 (18.3)

3. Primary Outcome: OZ439 C168h
Description: OZ439 concentration observed at 168h
Time Frame: 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2, Treatment B: Single Oral Dose of 800 mg OZ439 | Part 2, Treatment C: Single Oral Dose of 400 mg OZ439 | Part 2, Treatment D:Single Oral Dose 400 mg OZ439+Cobicistat
Number analyzed (Participants) | 18 | 18 | 18
ng/mL | 3.54 (65.3) | 2.48 (83.1) | 6.07 (46.6)

4. Primary Outcome: OZ439 AUC0-168h
Description: Area under the OZ439 plasma concentration time curve from time zero to 168h
Time Frame: Pre-dose, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Part 2, Treatment B: Single Oral Dose of 800 mg OZ439 | Part 2, Treatment C: Single Oral Dose of 400 mg OZ439 | Part 2, Treatment D:Single Oral Dose 400 mg OZ439+Cobicistat
Number analyzed (Participants) | 18 | 18 | 18
ng.h/mL | 9857 (37.3) | 6049 (51.5) | 13949 (25.6)

5. Primary Outcome: OZ439 AUC0-inf
Description: Area under the OZ439 plasma concentration time curve from time zero to infinity
Time Frame: Pre-dose, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 168, 216, 264, 312 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Part 2, Treatment B: Single Oral Dose of 800 mg OZ439 | Part 2, Treatment C: Single Oral Dose of 400 mg OZ439 | Part 2, Treatment D:Single Oral Dose 400 mg OZ439+Cobicistat
Number analyzed (Participants) | 18 | 18 | 18
ng.h/mL | 10222 (37.4) | 6378 (52.3) | 14984 (25.7)

ADVERSE EVENTS:
Time Frame: Day -28 (screening) to Day 15 (follow-up)
Description: 13 subjects (50%) reported a total of 29 TEAEs. In addition, a total of 3 AEs that had started prior to dosing were reported. These AEs did not preclude randomization and dosing of the subjects. There were no deaths or SAEs reported during the study. All TEAEs were transient and resolved without sequelae. One TEAE was still ongoing at the time of follow-up. None of the subjects were discontinued during the study due to TEAEs.
Groups:
- Part 1, Single Arm: This was an open-label study in 8 healthy subjects to determine the absolute bioavailability of OZ439 following a single oral dose of OZ439 and co-administration of a single iv infusion of a [14C]-OZ439 radiolabeled microdose at the anticipated Tmax of the oral dose. Subjects received the following treatment:
  Treatment A: A single oral dose of 800 mg OZ439 simple granules administered as a 100-mL dispersion followed by a 15-minute 10-mL iv infusion of 100 μg [14C]-OZ439 (47 kBq [1.27 μCi]) beginning 3 hours after the oral dose administration.
  Single oral dose of 800 mg OZ439: Single oral dose of 800 mg OZ439
  iv infusion of [14C]-OZ439: 15-minute 10-mL iv infusion of 100 μg [14C]-OZ439
Arm/Group | Part 1, Single Arm | Part 2, Treatment B: Single Oral Dose of 800 mg OZ439 | Part 2, Treatment C: Single Oral Dose of 400 mg OZ439 | Part 2, Treatment D:Single Oral Dose 400 mg OZ439+Cobicistat
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/8 | 10/18 | 4/18 | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Single Arm (N=8) | Part 2, Treatment B: Single Oral Dose of 800 mg OZ439 (N=18) | Part 2, Treatment C: Single Oral Dose of 400 mg OZ439 (N=18) | Part 2, Treatment D:Single Oral Dose 400 mg OZ439+Cobicistat (N=18)
Injection Site Irritation (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Feeling Cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection Site Haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysphonia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PRA shall have the right to publish the results of the research, subject to the sponsor's prior written consent, which shall not be unreasonably withheld or delayed. Following the receipt of such consent, PRA shall submit a copy of the proposed publication to the sponsor who shall have 30 days in which to request amendments thereto which, to the extent that such proposed amendments are reasonable, PRA shall be obliged to incorporate prior to such publication.

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT04069221/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT04069221/SAP_001.pdf